CLINICAL TRIAL: NCT04804449
Title: Prospective Longitudinal Effects of Intra-articular Corticosteroid Injection on Synovial Fluid Oxygen
Acronym: POLO
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 15303
Record Dates: First submitted 2021-03-08; First posted 2021-03-18 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid arthritis and psoriatic arthritis: Patients with rheumatoid arthritis or psoriatic arthritis, who require an intra-articular corticosteroid injection

SUMMARY:
Inflammatory arthritis such as rheumatoid arthritis (RA) and psoriatic arthritis (PsA) are characterized by synovial inflammation of joints, potentially leading to joint destruction and functional disability. Inflamed joints have lower oxygen levels. Studying how oxygen level within the joint affect inflammation may lead to new treatments for patients with arthritis. Anti-inflammatory corticosteroid injection into the joint is well tolerated and widely used in clinical practice but its effects on oxygen level within joints is unknown. Therefore, patients who require corticosteroid injection into the joint as routine clinical care will have biological samples collected before and after the injection. This will give new information to put into context the biological effects within the joint, and accelerate development of new treatment approaches in the future.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Fulfil American College of Rheumatology/European League Against Rheumatism criteria (ACR/EULAR) 2010 Rheumatoid Arthritis Classification Criteria or fulfil Classification Criteria for Psoriatic Arthritis 2006 (CASPAR).
* Participant has been selected for intra-articular corticosteroid injection as part of their routine clinical care.
* Selected joint for biopsy must be minimum Grade 2 synovial thickening for large joint (knee) and medium joint (wrist), or minimum Grade 3 synovial thickening for small joint (metacarpophalangeal).

Exclusion Criteria:

* Current enrolment in any other clinical study involving an investigational study treatment.
* Intramuscular, intravenous or intra-articular administration of corticosteroid within 4 weeks prior to baseline visit.
* Oral corticosteroid > 10 mg/day prednisolone or equivalent within 4 weeks prior to baseline visit.
* Oral corticosteroid dose not stable for at least 4 weeks prior to baseline visit.
* Oral non-steroidal anti-inflammatory drugs (including aspirin > 75 mg/ day and selective-cyclooxygenase inhibitors) dose not stable for at least 4 weeks prior to baseline visit.
* Disease modifying anti-rheumatic drugs (DMARDs) dose not stable for at least 4 weeks prior to baseline visit.
* History of septic arthritis.
* Participants on warfarin, heparin, low molecular weight heparin, direct oral anticoagulants. Oral anti-platelet agents are permitted.
* History of haemophilia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with rheumatoid arthritis or psoriatic arthritis who require intra-articular corticosteroid injection, and swollen joint suitable for ultrasound guided synovial biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Effects of intra-articular corticosteroid injection on joint oxygen tension in patients with rheumatoid and psoriatic arthritis | Day 28
  Change from Baseline Synovial fluid partial pressure of oxygen at Day 28

SECONDARY OUTCOMES:
Effects of intra-articular corticosteroid injection on joint hypoxia in patients with rheumatoid and psoriatic arthritis | Day 1 and 28
  Hypoxia-inducible factor 1α (HIF-1α) protein levels in synovial tissues
Effects of intra-articular corticosteroid injection on synovial fibroblast protein expression | Day 28
  Change from baseline protein expression levels in synovial fibroblasts at Day 28
Effects of intra-articular corticosteroid injection on patient satisfaction | Day 28
  Treatment Satisfaction Questionnaire (TSQM)©

CONTACTS AND LOCATIONS:
Overall Officials: Shing Law, BM BCh, Principal Investigator — University of Oxford
Locations (1):
- Nuffield Orthopaedic Centre, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No